CLINICAL TRIAL: NCT06393036
Title: The Effect of Obstructive Sleep Apnea on Severity and Prognosis of Patients With IgA Nephropathy
Brief Title: The Effect of OSA on Severity and Prognosis of Patients With IgAN
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xiaowan Du, Principal Investigator, Peking University First Hospital
Other Study IDs: PekingUFH ENT OSAIgAN V1.0
Record Dates: First submitted 2024-04-24; First posted 2024-05-01 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea; IgA Nephropathy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Glomerulonephritis, IGA | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients diagnosed with both OSA and IgAN: Patients diagnosed with both OSA and IgAN, and treated with CPAP in addition to nephrological drug therapy or not.
  Interventions: Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — The intervention in this study involves the use of Continuous Positive Airway Pressure (CPAP) treatment. Although the study is designed as an observational cohort study, where patients self-selected whether to receive treatment rather than being assigned, there is still an intervention project, CPAP, present in the observational cohort. CPAP is a commonly used therapy for obstructive sleep apnea (OSA) and other sleep-related breathing disorders. The principle of CPAP treatment lies in maintaining a constant airway pressure during sleep to prevent the collapse of the upper airway and ensure unobstructed breathing. The patient wears a mask connected to a CPAP machine, which generates a steady stream of air to provide the necessary pressure.

SUMMARY:
This study aims to investigate the influence of obstructive sleep apnea hypopnea syndrome (OSA) on the severity and prognosis of patients with IgA nephropathy (IgAN), and to evaluate the therapeutic effect of continuous positive airway pressure (CPAP) intervention in such patients. Although the study is designed as an observational cohort study, where patients self-selected whether to receive treatment rather than being assigned, there is still an intervention project, CPAP, present in the observational cohort. Through a cohort study design, scientific evidences are expected for clinical decision-making and optimize treatment strategies for patients with OSA and IgAN.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria: IgA nephropathy is diagnosed based on the pathological results of renal biopsy and/or clinical manifestations (such as hematuria, proteinuria, abnormal renal function, etc.), in accordance with the internationally recognized diagnostic criteria for IgA nephropathy. Obstructive sleep apnea-hypopnea syndrome (OSAHS) is confirmed through overnight polysomnography (PSG) with an apnea-hypopnea index (AHI) of ≥5 events per hour, primarily consisting of obstructive events.
* Age and gender: Participants must be ≥18 years old, with no gender restrictions (as both OSAHS and IgA nephropathy do not show significant gender predisposition).
* Informed consent: Participants are required to voluntarily sign a written informed consent form, acknowledging and agreeing to participate in the study, including all its contents and potential risks.

Exclusion Criteria:

* Other sleep-related breathing disorders: Participants with mixed sleep apnea, central sleep apnea, or severe snoring with an AHI index of <5 events per hour will be excluded to ensure that the study population is limited to patients with OSAHS.
* Severe internal medical conditions: Patients with severe cardiopulmonary dysfunction, malignancy, severe liver disease, mental disorders, or other severe internal medical conditions that may significantly affect sleep or the progression of kidney disease will be excluded.
* Recent surgery or medication: Individuals who have undergone surgery within the past 3 months that may affect sleep or kidney function, or who are currently using medications that may significantly interfere with sleep or the assessment of kidney disease (such as corticosteroids, immunosuppressants, novel antipsychotics, etc.) will be excluded.
* Pregnant women.
* Inability to cooperate with the study: Patients who are unable to complete the study procedures (including polysomnography, follow-up, etc.) due to cognitive impairment, language communication difficulties, remote residence, or other reasons will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with both OSA and IgAN
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | 2 years

SECONDARY OUTCOMES:
Rate of kidney failure | 5 years
Kidney dialysis rate | 5 years

OTHER OUTCOMES:
change in serum creatinine | 2 years
change in serum eGFR | 2 years
change in blood urea nitrogen | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowan Du, Study Director — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be provided upon request.